CLINICAL TRIAL: NCT05629273
Title: Long Term Renal Function After CRRT in the Paediatric Intensive Care Unit, a Follow-up Study.
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-01669-02
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury; Multi Organ Failure; Children, Only
Keywords: Acute kidney injury; Multi organ failure; Children; Long term complications; Chronic renal damage
MeSH Terms: conditions — Acute Kidney Injury; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children treated with continuous renal replacement therapy in the intensive care unit.: Children treated with CRRT in the ICU due to AKI stage ≥1 (according to KDIGO) and/or ≥2 organ failures. The aim is to evaluate their long term renal function and establish the frequency of chronic kidney disease. Nephrology follow up will be done by a pediatric nephrologist for children living in the Stockholm area or have ongoing care at Karolinska University Hospital.
  Due to high mortality in this group of patients and the fact that many patients are referred to Karolinska University Hospital from other regions in Sweden, a substantial number of patients will be lost to follow-up. The investigators will therefore conduct a register-based study of all children who received CRRT due to AKI and/or MOF at Karolinska University Hospital from 2008-2021. Data regarding mortality, cause of death and diagnosis of chronic renal disease will be collected from the Swedish National Patient Register and National Cause of Death Register.

SUMMARY:
In this study the investigators will evaluate the long-term renal function in children treated with continuous renal replacement therapy (CRRT) due to acute kidney injury (AKI) and multiple organ failure (MOF) in the pediatric intensive care unit (PICU). These children are not always referred for nephrology follow up after their ICU stay and it is unclear to what extent the patients suffer from chronic renal disease. The primary aim is to establish the frequency of chronic kidney disease (CKD) in children treated with CRRT due to AKI. Secondary outcomes will include mortality, frequency of end stage-renal disease (ESRD) and need for hemodialysis and/or renal transplantation.

DETAILED DESCRIPTION:
-Background: Children receiving CRRT due to AKI are a group of severely ill patients. The mortality is high, varying from 16-58 % in different studies (1). Degree of fluid overload at CRRT start is an independent risk factor for PICU mortality (2). MOF and low weight also contribute to a significantly increased mortality rate (3).

Previous studies on adults have shown that CRRT in the ICU is an independent risk factor for both in-hospital and long-term mortality, as well as the development of CKD and end-stage renal disease. Patients with continued impaired renal function at ICU discharge are at higher risk, but patients with complete recovery of their AKI are also at risk of adverse long-term outcomes (4). Data describing the incidence of chronic renal disease after pediatric CRRT are scarce.

Many pediatric ICU patients with AKI don´t have clinical signs of renal damage after ICU discharge (5-8). However, the kidneys do have a capacity to compensate for renal damage and subclinical decreased renal function is not always detected. Subclinical renal damage in children can over the years develop into more severe renal damage and significant symptoms may appear later in life. Recent data show that AKI in the pediatric ICU leads to increased long-term mortality as well as renal damage (5, 9, 10). However, these studies mainly include older children and also covers milder degrees of AKI. Studies investigating long term outcomes after pediatric CRRT are needed. Moreover, it is important to identify risk factors for the development of chronic renal disease in these children in order to initiate adequate follow up and preventive treatment.

-Methods: This is a combined retrospective and prospective single center observational cohort study. All pediatric patients treated with CRRT from 2008 to 2021 at Karolinska University Hospital in Stockholm will be evaluated for enrollment. Data regarding patient characteristics in the PICU and CRRT data will retrospectively be collected from their medical chart. These data include age and weight at CRRT initiation and hospital discharge, comorbidities, reason for ICU admission, mechanical ventilation and ECMO treatment. Data regarding renal function include CRRT indication, KDIGO and PELOD 2 stage at CRRT initiation, serum-creatinine, serum-chloride at CRRT initiation, serum-creatinine at PICU discharge, urine dipstick and urine-albumin/creatinine ratio.

For patients with no nephrology follow-up after CRRT treatment, the renal function will be evaluated by a pediatric nephrologist. Due to practical matters however, this is only possible for patients from the Stockholm area and patients with ongoing care at Karolinska University Hospital. Renal function will be evaluated using serum Creatinine and Cystatin C. Follow-up will also include urine dipstick, urine albumin/creatinine ratio and blood pressure. Further investigations, such as renal ultrasonography or scintigraphy will be performed if deemed clinically relevant. For patients that have already had nephrology follow-up after CRRT, data will be collected from patient charts.

A substantial number of patients will be lost to prospective follow-up due to the high mortality in this group of patients and the fact that many patients are referred to Karolinska University Hospital from other regions in Sweden.

In order to describe the mortality and the risk of symptomatic chronic renal disease after pediatric CRRT the investigators will also conduct a retrospective register-based study of all children who received CRRT due to AKI and/or CRRT at Karolinska University Hospital from 2008-2021. Data regarding mortality, cause of death and diagnosis of chronic renal disease will be collected from the Swedish National Patient Register and National Cause of Death Register. Patients referred from outside Sweden will be excluded from this part of the study.

ELIGIBILITY:
Inclusion Criteria:

- Age newborn to 18 when admitted to ICU. CRRT treatment 2008-2021 due to AKI stage ≥ stage 1 (according to KDIGO) and/or ≥ 2 organ failures

Exclusion Criteria:

* CRRT due to metabolic and/or endocrinologic comorbidity.
* Chronic renal failure before CRRT.
* Previous renal transplantation.

Prospective part:

- Not a resident of Stockholm County and no planned follow up at Karolinska University Hospital.

Retrospective part:

- Patient referred to Karolinska University Hospital from a hospital outside Sweden.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children treated with CRRT in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Chronic renal disease (CKD) | Up to12 years.
  Frequency of chronic renal disease (CKD) according to KDIGO definitions at nephrology follow-up.
Chronic renal disease (CKD) | Up to 12 years
  Frequency of chronic renal disease according to ICD diagnosis in Swedish National Patient Register.

SECONDARY OUTCOMES:
Hypertension | Up to 12 years
  Frequency of hypertension at nephrology follow-up.
End-stage renal disease | Up to 12 years
  Frequency of end-stage renal disease defined as the need for renal transplantation or dialysis at nephrology follow up.
Hypertension | Up to 12 years
  Frequency of hypertension according to ICD diagnosis in Swedish National Patient Register.
Dialysis Therapy. | Up to 12 years
  Frequency of dialysis therapy according to Swedish National Patient Register.
Renal transplantation | Up to 12 years
  Frequency of renal transplantation according to Swedish National Patient Register
Mortality | Up to 1 year
  PICU mortality
Mortality | Up to 12 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Urban Fläring, Principal Investigator — Children Perioperative Medicine & Intensive Care, Karolinska University Hospital
Locations (1):
- Pediatric Perioperative Medicine and Intensive Care, Stockholm, Sweden, Sweden

REFERENCES:
- [Background] Almarza S, Bialobrzeska K, Casellas MM, Santiago MJ, Lopez-Herce J, Toledo B, Carrillo A. [Long-term outcomes of children treated with continuous renal replacement therapy]. An Pediatr (Barc). 2015 Dec;83(6):404-9. doi: 10.1016/j.anpedi.2014.12.018. Epub 2015 Feb 13. Spanish. PMID 25683273
- [Background] Andersson A, Norberg A, Broman LM, Martensson J, Flaring U. Fluid balance after continuous renal replacement therapy initiation and outcome in paediatric multiple organ failure. Acta Anaesthesiol Scand. 2019 Sep;63(8):1028-1036. doi: 10.1111/aas.13389. Epub 2019 Jun 3. PMID 31157412
- [Background] Sutherland SM, Zappitelli M, Alexander SR, Chua AN, Brophy PD, Bunchman TE, Hackbarth R, Somers MJ, Baum M, Symons JM, Flores FX, Benfield M, Askenazi D, Chand D, Fortenberry JD, Mahan JD, McBryde K, Blowey D, Goldstein SL. Fluid overload and mortality in children receiving continuous renal replacement therapy: the prospective pediatric continuous renal replacement therapy registry. Am J Kidney Dis. 2010 Feb;55(2):316-25. doi: 10.1053/j.ajkd.2009.10.048. Epub 2009 Dec 30. PMID 20042260
- [Background] Wu L, Zhang P, Yang Y, Jiang H, He Y, Xu C, Yan H, Guo Q, Luo Q, Chen J. Long-term renal and overall survival of critically ill patients with acute renal injury who received continuous renal replacement therapy. Ren Fail. 2017 Nov;39(1):736-744. doi: 10.1080/0886022X.2017.1398667. PMID 29199512
- [Background] Askenazi DJ, Feig DI, Graham NM, Hui-Stickle S, Goldstein SL. 3-5 year longitudinal follow-up of pediatric patients after acute renal failure. Kidney Int. 2006 Jan;69(1):184-9. doi: 10.1038/sj.ki.5000032. PMID 16374442
- [Background] Hayes LW, Oster RA, Tofil NM, Tolwani AJ. Outcomes of critically ill children requiring continuous renal replacement therapy. J Crit Care. 2009 Sep;24(3):394-400. doi: 10.1016/j.jcrc.2008.12.017. Epub 2009 Mar 27. PMID 19327959
- [Background] Diane Mok TY, Tseng MH, Chiang MC, Lin JL, Chu SM, Hsu JF, Lien R. Renal replacement therapy in the neonatal intensive care unit. Pediatr Neonatol. 2018 Oct;59(5):474-480. doi: 10.1016/j.pedneo.2017.11.015. Epub 2017 Dec 21. PMID 29396136
- [Background] Morelli S, Ricci Z, Di Chiara L, Stazi GV, Polito A, Vitale V, Giorni C, Iacoella C, Picardo S. Renal replacement therapy in neonates with congenital heart disease. Contrib Nephrol. 2007;156:428-33. doi: 10.1159/000102134. PMID 17464154
- [Background] Calderon-Margalit R, Golan E, Twig G, Leiba A, Tzur D, Afek A, Skorecki K, Vivante A. History of Childhood Kidney Disease and Risk of Adult End-Stage Renal Disease. N Engl J Med. 2018 Feb 1;378(5):428-438. doi: 10.1056/NEJMoa1700993. PMID 29385364
- [Background] Mammen C, Al Abbas A, Skippen P, Nadel H, Levine D, Collet JP, Matsell DG. Long-term risk of CKD in children surviving episodes of acute kidney injury in the intensive care unit: a prospective cohort study. Am J Kidney Dis. 2012 Apr;59(4):523-30. doi: 10.1053/j.ajkd.2011.10.048. Epub 2011 Dec 28. PMID 22206744